CLINICAL TRIAL: NCT05228730
Title: A Randomised Controlled Trial to Assess the Immunogenicity, Safety, and Reactogenicity of Standard-dose Versus Fractional Doses of COVID-19 Vaccines (Pfizer-BioNTech or Moderna) Given as an Additional Dose After Priming With Pfizer-BioNTech or AstraZeneca in Healthy Adults in Australia-MIACoV
Brief Title: Evaluation of Full Versus Fractional Doses of COVID-19 Vaccines Given as a Booster in Adults in Australia - Mongolia, Indonesia, Australia Coronavirus (MIACoV).
Acronym: MIACoV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the small number of participants
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 81764
Record Dates: First submitted 2022-02-05; First posted 2022-02-08 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: Booster dose; Moderna; Pfizer; fractional and standard doses; COVID-19 vaccination; mRNA vaccine
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Study participants who have received two doses of either Pfizer or Astrazena vaccine as their primary vaccine will be randomised into one of four groups. The four groups consists of a standard or fractional dose of either Pfizer or Moderna vaccine.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and those evaluating reactogenicity will be blinded to the vaccine allocation for the first 28 days following vaccination. After that, both clinical investigators and participants will be aware of their investigational product allocation. Laboratory staff will remain blinded to the investigational product allocation during the immunology testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Standard Pfizer-BioNTech booster group (Active Comparator): Received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine
  Interventions: Biological: Tozinameran - Standard dose
- Fractional Pfizer-BioNTech booster group (Experimental): Received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine
  Interventions: Biological: Tozinameran - fractional dose
- Standard Elasomeran booster group (Active Comparator): Received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine
  Interventions: Biological: Elasomeran - standard dose
- Fractional Elasomeran booster group (Experimental): Received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine
  Interventions: Biological: Elasomeran - fractional dose

INTERVENTIONS:
Biological: Tozinameran - Standard dose — Tozinamrean is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS_CoV-2). A standard dose will be administered on day 0 of the study.
  Other Names: BNT162b2; Pfizer-BioNTech; Comirnaty
  Arms: Standard Pfizer-BioNTech booster group
Biological: Tozinameran - fractional dose — Tozinamrean is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS_CoV-2). A fractional dose (15mcg) of the intervention will be administered on day 0 of the study.
  Other Names: BNT162b2; Comirnaty; Pfizer-BioNTech
  Arms: Fractional Pfizer-BioNTech booster group
Biological: Elasomeran - standard dose — Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  A single standard dose (50mcg) of the intervention will be administered on day 0 of the study.
  Other Names: mRNA-1273; Spikevax; Moderna
  Arms: Standard Elasomeran booster group
Biological: Elasomeran - fractional dose — Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  A fractional dose (20mcg) of the intervention will be administered on day 0 of the study.
  Other Names: mRNA-1273; Spikevax; Moderna
  Arms: Fractional Elasomeran booster group

SUMMARY:
This is a single-blind, randomised controlled clinical trial to determine the reactogenicity and immunogenicity of severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) vaccines (Pfizer-BioNTech or Moderna) as booster dose in adults, who have previously received either Pfizer-BioNTech or AstraZeneca as their primary doses.

Both fractional and standard doses of Pfizer-BioNTech or Moderna will be tested.

The trial intervention will be given in line with Australian Technical Advisory Group on Immunisation (ATAGI) recommendations for booster vaccine doses which allows booster doses from 5 months onwards . There will be a total of 8 groups, with 100 individuals of even spread of participants above and below 50 years in each group. The trial will be single site, based at Royal Children's Hospital, Melbourne, Australia

DETAILED DESCRIPTION:
As per brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Have completed two doses of Pfizer-BioNTech or AstraZeneca vaccines with the recommended schedule 6 months prior to the date of enrolment
2. Willing and able to give written informed consent
3. Aged 18 years or above
4. Willing to complete the follow-up requirements of the study

Exclusion Criteria:

1. Received 3 doses of COVID-19 vaccine
2. Received 2 doses of COVID-19 less than 6 months prior to the start of the trial
3. Received a different Covid-19 vaccine not available in Australia
4. Currently on immunosuppressive medication or anti-cancer chemotherapy
5. HIV infection
6. Congenital immune deficiency syndrome
7. Has received immunoglobulin or other blood products in the 3 months prior to vaccination
8. Study staff and their relatives
9. Have a history of a severe allergic reaction to any COVID-19 vaccines or have a medical exception to receiving further COVID-19 vaccines
10. Cannot read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mulholland, MD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data to ethically approved studies in cases where participants have indicated on the consent form that they consent to the use of their data and where consistent with terms of collaboration agreements.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) sharing plans in development
Access Criteria: IPD sharing plans in development

REFERENCES:
- [Background] Munro APS, Janani L, Cornelius V, Aley PK, Babbage G, Baxter D, Bula M, Cathie K, Chatterjee K, Dodd K, Enever Y, Gokani K, Goodman AL, Green CA, Harndahl L, Haughney J, Hicks A, van der Klaauw AA, Kwok J, Lambe T, Libri V, Llewelyn MJ, McGregor AC, Minassian AM, Moore P, Mughal M, Mujadidi YF, Murira J, Osanlou O, Osanlou R, Owens DR, Pacurar M, Palfreeman A, Pan D, Rampling T, Regan K, Saich S, Salkeld J, Saralaya D, Sharma S, Sheridan R, Sturdy A, Thomson EC, Todd S, Twelves C, Read RC, Charlton S, Hallis B, Ramsay M, Andrews N, Nguyen-Van-Tam JS, Snape MD, Liu X, Faust SN; COV-BOOST study group. Safety and immunogenicity of seven COVID-19 vaccines as a third dose (booster) following two doses of ChAdOx1 nCov-19 or BNT162b2 in the UK (COV-BOOST): a blinded, multicentre, randomised, controlled, phase 2 trial. Lancet. 2021 Dec 18;398(10318):2258-2276. doi: 10.1016/S0140-6736(21)02717-3. Epub 2021 Dec 2. PMID 34863358
- See also: Quarter-dose of Moderna COVID vaccine still rouses a big immune response — https://www.nature.com/articles/d41586-021-01893-0
- See also: US Food and Drug Administration (FDA). Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials 2007 — https://www.fda.gov/media/73679/download

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were randomised and assigned to one of the eight groups. However, due to the small number of participants enrolled, we have combined the groups based on the vaccine they received during the study and not stratify based on their previous vaccination history.
Groups:
- Standard Elasomeran Booster Group: Received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine
  Elasomeran - standard dose: Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  A single standard dose (50mcg) of the intervention will be administered on day 0 of the study.
- Fractional Elasomeran Booster Group: Received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine
  Elasomeran - fractional dose: Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  A fractional dose (20mcg) of the intervention will be administered on day 0 of the study.
Period: Overall Study
Arm/Group | Standard Pfizer-BioNTech Booster Group | Fractional Pfizer-BioNTech Booster Group | Standard Elasomeran Booster Group | Fractional Elasomeran Booster Group
Started | 4 | 1 | 4 | 4
Completed | 4 | 1 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Pfizer-BioNTech Booster Group: Due to the small number of participants enrolled, we have combined the groups based on the vaccine they received (i.e. Standard Pfizer-BioNTech booster group) and did not stratify based on their previous vaccination history (i.e. received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
  Tozinameran - Standard dose: Tozinamrean is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS_CoV-2). A standard dose will be administered on day 0 of the study.
- Fractional Pfizer-BioNTech Booster Group: Due to the small number of participants enrolled, we have combined the groups based on the vaccine they received (i.e. fractional Pfizer-BioNTech booster group) and did not stratify based on their previous vaccination history (i.e. received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
  Tozinameran - fractional dose: Tozinamrean is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS_CoV-2). A fractional dose (15mcg) of the intervention will be administered on day 0 of the study.
- Standard Elasomeran Booster Group: Due to the small number of participants enrolled, we have combined the groups based on the vaccine they received (i.e. standard Elasomeran booster group) and did not stratify based on their previous vaccination history (i.e. received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
  Elasomeran - standard dose: Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  A single standard dose (50mcg) of the intervention will be administered on day 0 of the study.
- Fractional Elasomeran Booster Group: Due to the small number of participants enrolled, we have combined the groups based on the vaccine they received (i.e. fractional Elasomeran booster group) and did not stratify based on their previous vaccination history (i.e. received two doses of AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
  Elasomeran - fractional dose: Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  A fractional dose (20mcg) of the intervention will be administered on day 0 of the study.
- Total: Total of all reporting groups
Arm/Group | Standard Pfizer-BioNTech Booster Group | Fractional Pfizer-BioNTech Booster Group | Standard Elasomeran Booster Group | Fractional Elasomeran Booster Group | Total
Number analyzed (Participants) | 4 | 1 | 4 | 4 | 13
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 55.23 [35.6 to 68.1] | 33.5 [33.5 to 33.5] | 44.7 [44.7 to 51.7] | 40.6 [29.1 to 50.8] | 44.7 [33.5 to 51.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 3
  Male | 4 | 1 | 2 | 3 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Australian | 2 | 1 | 2 | 3 | 8
  Filipino | 1 | 0 | 0 | 0 | 1
  Korean | 1 | 0 | 1 | 0 | 2
  Polish | 0 | 0 | 0 | 1 | 1
  Serbian | 0 | 0 | 1 | 0 | 1
  Southern and East African | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 4 | 1 | 4 | 4 | 13
Any reaction to primary vaccine [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 2 | 2 | 6
  No | 2 | 1 | 2 | 2 | 7
Medical status at enrolment [Count of Participants; unit: Participants]
  *Gestational diabetes (female only) | 0 | 0 | 0 | 1 | 1
  *Pregnant (female only) | 0 | 0 | 1 | 0 | 1
  Cardiovascular disease | 0 | 0 | 1 | 0 | 1
  Cigarette use | 1 | 0 | 0 | 0 | 1
  Anticoagulant therapy | 0 | 0 | 2 | 0 | 2
Currently taking medication [Count of Participants; unit: Participants]
  No | 2 | 0 | 2 | 4 | 8
  Yes | 2 | 1 | 2 | 0 | 5
Ever tested positive to SARS-CoV-2 [Count of Participants; unit: Participants] | 0 | 1 | 2 | 4 | 7
Symptoms consistent with COVID-19 [Count of Participants; unit: Participants] | 0 | 1 | 2 | 4 | 7
Worst clinical spectrum of COVID-19 [Count of Participants; unit: Participants]
  Mild | 0 | 1 | 1 | 3 | 5
  Moderate | 0 | 0 | 1 | 1 | 2
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 25.5 [22 to 31.1] | 21.9 [21.9 to 21.9] | 27.8 [23.2 to 30.5] | 23.0 [21.5 to 24.6] | 24.4 [21.6 to 26.9]
Temperature [Median (Inter-Quartile Range); unit: celsius] | 36.3 [35.2 to 36.4] | 36.2 [36.2 to 36.2] | 35.9 [35.4 to 36.3] | 35.5 [35.5 to 35.6] | 35.7 [35.4 to 36.3]
Pulse rate pre COVID-19 booster dose [Median (Inter-Quartile Range); unit: beats/min] | 75 [68 to 81] | 66 [66 to 66] | 66 [56 to 80] | 71 [63 to 76] | 67 [65 to 76]
Respiratory rate pre COVID-19 booster dose [Median (Inter-Quartile Range); unit: breaths/min] | 17 [15 to 21] | 20 [20 to 20] | 14 [14 to 16] | 15 [13 to 18] | 16 [14 to 21]
Blood pressure pre- COVID-19 booster dose [Median (Inter-Quartile Range); unit: mmHG]
  Systolic | 125 [115.5 to 132] | 111 [111 to 111] | 119.5 [111.5 to 122] | 108 [99 to 109] | 111 [108 to 121]
  Diastolic | 83 [78.5 to 88] | 76 [76 to 76] | 75 [71 to 80.5] | 73.5 [68.5 to 82] | 76 [74 to 83]

OUTCOME MEASURES:

1. Primary Outcome: SARS-CoV-2 Specific Immunoglobulin (Ig)G Antibodies at 28-days Post Booster Vaccination
Description: Serum samples collected at 28-days post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using the commercial Euroimmun S1 IgG ELISA. Data will be reported as binding antibody units/mL and presented as geometric mean concentration and 95% confidence intervals
Time Frame: 28-days post booster vaccination.
Population: IgG antibody response 28-days post booster
Measure: Median (Inter-Quartile Range); unit: binding antibody units (BAU/mL)
Groups:
- Standard Pfizer-BioNTech Booster Group: Due to the small enrolment numbers in each group, we have combined the groups based on the vaccine that they received (Standard Pfizer-BioNTech) instead of stratifying the groups based on their previous vaccines received e.g. AstraZeneca or Pfizer).
- Fractional Pfizer-BioNTech Booster Group: Due to the small enrolment numbers in each group, we have combined the groups based on the vaccine that they received (Fractional Pfizer-BioNTech) instead of stratifying the groups based on their previous vaccines received e.g. AstraZeneca or Pfizer).
- Standard Elasomeran Booster Group: Due to the small enrolment numbers in each group, we have combined the groups based on the vaccine that they received (Standard Elasomeran) instead of stratifying the groups based on their previous vaccines received e.g. AstraZeneca or Pfizer).
- Fractional Elasomeran Booster Group: Due to the small enrolment numbers in each group, we have combined the groups based on the vaccine that they received (Fractional Elasomeran) instead of stratifying the groups based on their previous vaccines received e.g. AstraZeneca or Pfizer).
Arm/Group | Standard Pfizer-BioNTech Booster Group | Fractional Pfizer-BioNTech Booster Group | Standard Elasomeran Booster Group | Fractional Elasomeran Booster Group
Number analyzed (Participants) | 4 | 1 | 4 | 4
binding antibody units (BAU/mL) | 1927.1 [1665.4 to 3043.5] | 13707.2 [13707.2 to 13707.2] | 5118.6 [3837.6 to 8756.9] | 5908.7 [4926 to 6741.3]

ADVERSE EVENTS:
Time Frame: 7 days post vaccination
Description: Any untoward medical occurrence in a patient or clinical trial participant administered a medicinal product and does not necessarily have a causal relationship with this treatment.
Groups:
- Standard Pfizer-BioNTech Booster Group: Due to the low enrolment numbers, the groups were combined based on the vaccine they received (Standard Pfizer-BioNTech) and not stratified based on their vaccination history (AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
- Fractional Pfizer-BioNTech Booster Group: Due to the low enrolment numbers, the groups were combined based on the vaccine they received (Fractional Pfizer-BioNTech) and not stratified based on their vaccination history (AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
- Standard Elasomeran Booster Group: Due to the low enrolment numbers, the groups were combined based on the vaccine they received (Standard Elasomeran) and not stratified based on their vaccination history (AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
- Fractional Elasomeran Booster Group: Due to the low enrolment numbers, the groups were combined based on the vaccine they received (Fractional Elasomeran) and not stratified based on their vaccination history (AstraZeneca or Pfizer-BioNTech as primary COVID-19 vaccine).
Arm/Group | Standard Pfizer-BioNTech Booster Group | Fractional Pfizer-BioNTech Booster Group | Standard Elasomeran Booster Group | Fractional Elasomeran Booster Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/1 | 1/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Pfizer-BioNTech Booster Group (N=4) | Fractional Pfizer-BioNTech Booster Group (N=1) | Standard Elasomeran Booster Group (N=4) | Fractional Elasomeran Booster Group (N=4)
Throat infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tiredness (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrolment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT05228730/Prot_SAP_001.pdf